CLINICAL TRIAL: NCT00793793
Title: Safety, Antiviral Activity, and Pharmacokinetics of Multiple Rising Oral Doses of BI 201335 NA in Treatment-naïve Patients With Chronic Hepatitis C Infection for 14 Days Monotherapy Followed by Combination With Pegylated Interferon and Ribavirin for an Additional 14 Days (Double-blind, Placebo Controlled), and in Treatment-experienced Patients With Chronic Hepatitis C Infection for 28 Days as Combination Therapy With Pegylated Interferon and Ribavirin (Open-label)
Brief Title: Safety, Antiviral Activity and PK of MRD of BI 201335 in Chronic Hepatitis C Patients Both Treatment Naive and -Experienced
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.2; 2007-001158-19 (EudraCT Number)
Record Dates: First submitted 2008-09-23; First posted 2008-11-19 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir

ARMS (5):
- 20mg (Experimental): patient to receive 20mg solution BI201335 qd +/- PegIFN/RBV fore 28 days
  Interventions: Drug: BI201335
- 48mg (Experimental): patient to receive 48mg solution BI201335 qd +/- PegIFN/RBV fore 28 days
  Interventions: Drug: BI201335
- 120mg (Experimental): patient to receive 120mg solution BI201335 qd +/- PegIFN/RBV fore 28 days
  Interventions: Drug: BI201335
- 240mg (Experimental): patient to receive 240mg solution BI201335 qd +/- PegIFN/RBV fore 28 days
  Interventions: Drug: BI201335
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI201335 — patient to receive rising doses of BI201335 solution qd +/- PegIFN/RBV fore 28 days
  Arms: 240mg
Drug: BI201335 — patient to receive rising doses of BI201335 solution qd +/- PegIFN/RBV fore 28 days
  Arms: 120mg
Drug: BI201335 — patient to receive rising doses of BI201335 solution qd +/- PegIFN/RBV fore 28 days
  Arms: 48mg
Drug: BI201335 — patient to receive 240mg solution BI201335 qd +/- PegIFN/RBV fore 28 days
  Arms: 20mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate safety, antiviral activity, and pharmacokinetics of BI 201335 NA in HCV genotype 1 infected patients treated for 14 days monotherapy followed by BI 201335 NA combination therapy with PegIFN/RBV for an additional 14 days for treatment-naïve patients; or for 28 days as BI 201335 NA combination therapy with PegIFN/RBV for treatment-experienced patients.

A secondary objective is to investigate antiviral activity, potential drug-drug interactions and safety of combination therapy of BI 201335 NA and PegIFN/RBV up to 28 days for treatment-naïve patients.

ELIGIBILITY:
Inclusion criteria:

1a. For treatment-naïve patients: no prior therapy with interferon, peginterferon, or ribavirin for acute or chronic hepatitis C infection

1b. For treatment-experienced patients: confirmed virological failure during or after combination treatment with an approved dose of alfa-2a or alfa-2b peginterferon combined with ribavirin; such patients must have received at least 12 weeks of therapy with a 90 day washout period prior to screening and must have documentation of medical history prior to enrolment in 1220.2 2. Age 18 years or older 3. Signed informed consent form prior to trial participation 4. Male or female with documented hysterectomy or menopausal female with last menstrual period at least 6 months prior to screening 5. Chronic hepatitis C infection of genotype 1, diagnosed by positive HCV serology test (HCV Ab positive) or detectable HCV RNA at least 6 months prior to screening 6. HCV viral load >= 100,000 IU/mL at screening 7. TSH and T4 within normal limits or adequately controlled thyroid function 8. Histological evidence within 36 months prior to study enrolment of any degree of chronic necroinflammatory activity or the presence of fibrosis (Ishak Grade 1-4 or Metavir Grade 1-3)

Exclusion criteria:

1. Patients who have been previously treated with at least one dose of any protease inhibitor for acute or chronic hepatitis C infection
2. Evidence of liver disease due to causes other than chronic HCV infection
3. Positive ELISA for HIV-1 or HIV-2
4. Hepatitis B virus (HBV) infection based on presence of Hbs Ag or HBV DNA
5. Any previous liver biopsy consistent with cirrhosis
6. Decompensated liver diseases as evidenced by ascites, portal hypertension, jaundice or hepatic encephalopathy
7. Haemophilia
8. Hemoglobinopathy (e.g., thalassemia major or sickle cell anemia)
9. Severe pre-existing psychiatric disease
10. Poorly controlled diabetes mellitus
11. Ischaemic heart disease
12. Chronic obstructive airway disease
13. Autoimmune disease; including autoimmune hepatitis
14. History of alcohol abuse within the past 12 months
15. Hyperbilirubinemia (conjugated bilirubin) >1.5x ULN
16. Alkaline phosphatase >1.5x ULN
17. ALT and AST levels >= 5 x ULN
18. Hemoglobin < 12.0 g/dL for women and < 13.0 g/dL for men
19. White blood cell count < 2000 cells/mm3
20. Absolute Neutrophil Count < 1500 cells/mm3
21. Platelet count < 100,000 cells/mm3
22. Prothrombin time INR (Institutional Normalized Ratio) prolonged to > 1.5 x ULN
23. Usage of any investigational drug within 30 days prior to enrolment; or the planned usage of an investigational drug during the course of the current study
24. Known hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (16):
- United States (6):
  - 1220.2.10 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.2.15 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.2.17 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1220.2.11 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.2.12 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.2.14 Boehringer Ingelheim Investigational Site, Austin, Texas
- France (4):
  - 1220.2.3304A Boehringer Ingelheim Investigational Site, Lyon
  - 1220.2.3303A Boehringer Ingelheim Investigational Site, Marseille
  - 1220.2.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1220.2.3302A Boehringer Ingelheim Investigational Site, Paris
- Germany (5):
  - 1220.2.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.2.49005 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.2.49006 Boehringer Ingelheim Investigational Site, Hanover
  - 1220.2.49004 Boehringer Ingelheim Investigational Site, Kiel
  - 1220.2.49003 Boehringer Ingelheim Investigational Site, Mainz
- 1220.2.34001 Boehringer Ingelheim Investigational Site, Madrid, Spain

REFERENCES:
- [Derived] Berger KL, Lagace L, Triki I, Cartier M, Marquis M, Lawetz C, Bethell R, Scherer J, Kukolj G. Viral resistance in hepatitis C virus genotype 1-infected patients receiving the NS3 protease inhibitor Faldaprevir (BI 201335) in a phase 1b multiple-rising-dose study. Antimicrob Agents Chemother. 2013 Oct;57(10):4928-36. doi: 10.1128/AAC.00822-13. Epub 2013 Jul 22. PMID 23877706
- [Derived] Manns MP, Bourliere M, Benhamou Y, Pol S, Bonacini M, Trepo C, Wright D, Berg T, Calleja JL, White PW, Stern JO, Steinmann G, Yong CL, Kukolj G, Scherer J, Boecher WO. Potency, safety, and pharmacokinetics of the NS3/4A protease inhibitor BI201335 in patients with chronic HCV genotype-1 infection. J Hepatol. 2011 Jun;54(6):1114-22. doi: 10.1016/j.jhep.2010.08.040. Epub 2010 Nov 11. PMID 21145839

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Naive (TN): Placebo: TN patient to receive Placebo +/- Pegylated interferon alpha-2a solution for injection/Ribavirin tablet (PegIFN/RBV) for 28 days
- Treatment Naive(TN): 20mg Per Day (QD): TN patient to receive 20mg QD solution Faldaprevir (BI201335) qd +/- PegIFN/RBV for 28 days
- TN: 48mg QD: TN patient to receive 48mg solution BI201335 qd +/- PegIFN/RBV for 28 days
- TN: 120mg QD: TN patient to receive 120mg solution BI201335 qd +/- PegIFN/RBV for 28 days
- TN: 240mg QD: TN patient to receive 240mg solution BI201335 qd +/- PegIFN/RBV for 28 days
- Treatment Experienced (TE) Non-cirrhotic: 48 mg QD: TE non-cirrhotic patient to receive 48mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE Non-cirrhotic: 120 mg QD: TE non-cirrhotic patient to receive 120mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE Non-cirrhotic: 240 mg QD: TE non-cirrhotic patient to receive 240mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC): TE non-cirrhotic patient to receive 240mg QD SGC solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE Non-cirrhotic: 240 mg Twice a Day (BID) SGC: TE non-cirrhotic patient to receive 240mg BID SGC solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE With Cirrhosis: 240 mg QD SGC: TE with cirrhotic patient to receive 240mg QD SGC solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE With Cirrhosis: 240 mg BID SGC: TE with cirrhotic patient to receive 240mg BID SGC solution BI201335 qd +/- PegIFN/RBV for 28 days
Period: Overall Study
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg Twice a Day (BID) SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Started | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
Completed | 8 | 5 | 5 | 4 | 4 | 4 | 3 | 6 | 6 | 6 | 3 | 1
Not Completed | 0 | 1 | 2 | 3 | 2 | 2 | 4 | 0 | 9 | 9 | 3 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — reason not specified | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 7 | 6 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized patients who were dispensed trial medication and were documented to have taken at least 1 dose of trial medication.
Groups:
- Treatment Naive (TN): Placebo: TN patient to receive Placebo + PegIFN/RBV for 28 days
- TN: 20mg QD: TN patient to receive 20mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
- TE Non-cirrhotic: 240 mg BID SGC: TE non-cirrhotic patient to receive 240mg BID SGC solution BI201335 qd +/- PegIFN/RBV for 28 days
- Total: Total of all reporting groups
Arm/Group | Treatment Naive (TN): Placebo | TN: 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC | Total
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.88 (8.36) | 51.00 (7.97) | 47.14 (13.84) | 48.57 (16.31) | 47.83 (9.26) | 46.83 (11.82) | 46.71 (4.79) | 49.33 (10.11) | 50.93 (8.13) | 48.93 (13.10) | 53.67 (5.32) | 53.57 (8.36) | 49.59 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 1 | 2 | 3 | 3 | 5 | 7 | 1 | 2 | 30
  Male | 6 | 6 | 5 | 5 | 5 | 4 | 4 | 3 | 10 | 8 | 5 | 5 | 66

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: VR (Virologic Response) of >=2 log10 Reduction in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) From Baseline at Any Time up to Day 14 (naïve Patients) or Day 28 (Experienced Patients)
Description: Efficacy endpoint: VR (virologic response) of >=2 log10 reduction in Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) from baseline at any time up to Day 14 (naïve patients) or Day 28 (experienced patients).
Time Frame: Baseline and up to 4 weeks
Population: Full Analysis Set (FAS): All randomized TN patients and treatment experienced patients who were dispensed trial medication and were documented to have taken at least 1 dose of trial medication.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- TN: Placebo: TN patient to receive Placebo +/- PegIFN/RBV for 28 days
- Treatment Naive(TN): 20mg QD: TN patient to receive 20mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.00 [0.000 to 33.627] | 83.33 [42.128 to 96.331] | 100.00 [63.058 to 100.000] | 100.00 [63.058 to 100.000] | 100.00 [59.038 to 100.000] | 100.00 [59.038 to 100.000] | 100.00 [63.058 to 100.000] | 100.00 [59.038 to 100.000] | 100.00 [79.409 to 100.000] | 100.00 [79.409 to 100.000] | 100.00 [59.038 to 100.000] | 100.00 [63.058 to 100.000]

2. Primary Outcome: Occurrence of Adverse Events (AEs) During BI201335 + Washout Period
Description: Occurrence of Adverse Events (AEs) during BI201335 + washout period. For placebo patients include all AEs through 30 days after trial discontinuation.
Time Frame: from day 1 and up to 4 weeks + 4 days washout
Population: Treated Set (TS): This patient set included all patients who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment regardless of randomization.
Measure: Number; unit: percentage of participants with AEs
Groups:
- Treatment Experienced (TE) Non-cirrhotic: 48 mg QD: TE non-cirrhotic patient to receive 48 mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants with AEs | 62.5 | 100.0 | 100.0 | 57.1 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Primary Outcome: Occurrence of Serious Adverse Events (SAEs) During BI201335 + Washout Period
Description: Occurrence of Serious Adverse Events (SAEs)during BI201335 or BI201335+ washout period. For placebo patients include all SAEs through 30 days after trial discontinuation.
Time Frame: from day 1 and up to 4 weeks + 4 days washout
Population: TS
Measure: Number; unit: percentage of participants with SAEs
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants with SAEs | 0.0 | 16.7 | 14.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 28.6

4. Primary Outcome: Occurrence of Laboratory Test Abnormalities and With Respect to Division of AIDS (DAIDS) Classification and Laboratory Test Values Change Over Time
Description: Occurrence of laboratory test abnormalities and with respect to Division of AIDS (DAIDS) classification and laboratory test values change over time.
  ALT=Alanine transaminase (SGPT), AST=Aspartate transaminase (SGOT).
Time Frame: Baseline and up to 4 weeks
Population: TS
Measure: Number; unit: participants with grade 3 or 4 abnormal
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
participants with grade 3 or 4 abnormal
  ALT/GPT SGPT increase, with grade 3 or 4 abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AST/GOT SGOT increase, with grade 3 or 4 abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Lipase increase, with grade 3 or 4 abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Bilirubin total increa, with grade 3 or 4 abnormal | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 8 | 12 | 5 | 5
  Uric acid increase, with grade 3 or 4 abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Triglyceride increase, with grade 3 or 4 abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

5. Secondary Outcome: Maximum Viral Load Reduction From Baseline up to Day 14 for Treatment-naïve Patients and Day 28 Treatment for Treatment-experienced Patients
Description: Maximum viral load reduction from baseline up to Day 14 for treatment-naïve patients and Day 28 treatment for treatment-experienced patients.
Time Frame: Baseline and up to 4 weeks
Population: FAS (as randomised)
Measure: Median (Inter-Quartile Range); unit: log10 IU/mL
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
log10 IU/mL | -0.060 [-0.216 to 0.012] | -3.049 [-3.376 to -2.181] | -3.624 [-3.744 to -3.359] | -3.740 [-3.869 to -3.426] | -4.413 [-4.438 to -3.943] | -5.023 [-5.150 to -4.342] | -5.244 [-5.796 to -4.035] | -5.334 [-5.692 to -4.916] | -5.246 [-5.621 to -5.133] | -5.404 [-5.469 to -4.936] | -4.841 [-5.322 to -4.763] | -5.476 [-5.544 to -3.853]

6. Secondary Outcome: Change From Baseline in Viral Load on Day 14 for Treatment-naïve Patients and on Day 28 Treatment for Treatment-experienced Patients
Description: Change from baseline in viral load on Day 14 for treatment-naïve patients and on Day 28 treatment for treatment-experienced patients.
Time Frame: Baseline and up to 4 weeks
Population: FAS (as randomised) including patients with available viral load data.
Measure: Median (Inter-Quartile Range); unit: Log10 IU/mL
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 5 | 15 | 15 | 6 | 6
Log10 IU/mL | 0.209 [0.165 to 0.321] | -1.226 [-1.492 to -0.831] | -1.539 [-2.885 to -0.782] | -0.781 [-1.967 to -0.046] | -2.449 [-3.502 to -1.360] | -5.023 [-5.150 to -3.049] | -5.244 [-5.800 to -4.035] | -5.386 [-5.692 to -5.283] | -5.246 [-5.621 to -5.133] | -5.404 [-5.469 to -4.797] | -4.782 [-5.322 to -4.628] | -5.497 [-5.544 to -5.300]

7. Secondary Outcome: Rapid Virologic Response (RVR)
Description: Rapid virologic response (RVR): Plasma HCV RNA level below the limit of detection of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) on Day 28 for all patients.
Time Frame: week 4
Population: FAS (as randomized)
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.00 [0.000 to 33.627] | 0.00 [0.000 to 40.962] | 28.57 [8.523 to 65.086] | 14.29 [3.185 to 52.651] | 16.67 [3.669 to 57.872] | 33.33 [9.899 to 70.958] | 14.29 [3.185 to 52.651] | 16.67 [3.669 to 57.872] | 26.67 [11.017 to 52.377] | 26.67 [11.017 to 52.377] | 66.67 [29.042 to 90.101] | 14.29 [3.185 to 52.651]

8. Secondary Outcome: Early Virologic Response (EVR)
Description: Early Virologic Response (EVR): >=2 log10 reduction in plasma HCV RNA level from baseline at week 12 (day 84)
Time Frame: week 12
Population: FAS
Measure: Number; unit: percentage of responders
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.0 | 100.0 | 100.0 | 85.7 | 83.3 | 83.3 | 71.4 | 100.0 | 86.7 | 86.7 | 100.0 | 71.4

9. Secondary Outcome: Complete EVR1 (cEVR1)
Description: VL (Viral load) below the limit of quantification of the Roche COBAS Taqman HCV/HPS assay (25 IU/mL) at 4 weeks and below the limit of detection of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) at 12 weeks
Time Frame: week 4 and week 12
Population: FAS
Measure: Number; unit: percentage of responders
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.0 | 16.7 | 28.6 | 28.6 | 50.0 | 50.0 | 57.1 | 83.3 | 53.3 | 60.0 | 83.3 | 57.1

10. Secondary Outcome: Complete EVR2 (cEVR2)
Description: VL below the limit of detection at both 4 weeks and 12 weeks
Time Frame: week 4 and week 12
Population: FAS
Measure: Number; unit: percentage of responders
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.0 | 0.0 | 28.6 | 14.3 | 33.3 | 50.0 | 14.3 | 16.7 | 33.3 | 20.0 | 33.3 | 28.6

11. Secondary Outcome: End of Treatment Response (ETR)
Description: End of Treatment Response (ETR): Plasma HCV RNA level below the limit of detection of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) at week 48 (Day 336).
Time Frame: week 48
Population: FAS
Measure: Number; unit: percentage of responders
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.0 | 83.3 | 57.1 | 57.1 | 66.7 | 33.3 | 57.1 | 66.7 | 53.3 | 40.0 | 50.0 | 14.3

12. Secondary Outcome: Sustained Virologic Response (SVR)
Description: Sustained Virologic Response (SVR): Plasma HCV RNA level below the limit of detection of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) at week 72 (Day 504).
Time Frame: week 72
Population: FAS
Measure: Number; unit: percentage of responders
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of responders | 0.0 | 50.0 | 42.9 | 42.9 | 50.0 | 50.0 | 42.9 | 50.0 | 46.7 | 40.0 | 50.0 | 14.3

13. Secondary Outcome: Achievement of an HCV RNA Level Below the Limit of Detection Over Time
Description: Achievement of an HCV RNA level below the limit of detection of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) over time
Time Frame: from day 1 and up to 4 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Groups:
- TN: Placebo: TN patient to receive Placebo +/- Pegylated interferon alpha-2a solution for injection/Ribavirin tablet (PegIFN/RBV) for 28 days
- Treatment Naive(TN): 20mg QD: TN patient to receive 20mg QD solution Faldaprevir (BI201335) qd +/- PegIFN/RBV for 28 days
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg BID SGC | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants | 0.0 | 0.0 | 28.6 | 14.3 | 16.7 | 33.3 | 14.3 | 16.7 | 26.7 | 26.7 | 66.7 | 14.3

14. Secondary Outcome: Achievement of an HCV RNA Level Below the Limit of Quantification Over Time
Description: Achievement of an HCV RNA Level Below the Limit of quantification of the Roche COBAS Taqman HCV/HPS assay (25 IU/mL) Over Time
Time Frame: from day 1 and up to 4 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg BID SGC | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants | 0.0 | 16.7 | 28.6 | 28.6 | 50.0 | 50.0 | 57.1 | 83.3 | 66.7 | 60.0 | 83.3 | 85.7

15. Secondary Outcome: Achievement of a >= 2 log10 Reduction in Plasma HCV RNA Level From Baseline Over Time
Description: Achievement of a >= 2 log10 reduction in plasma HCV RNA level from baseline over time.
Time Frame: from day 1 and up to 4 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg BID SGC | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants | 0.0 | 83.3 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

16. Secondary Outcome: Occurrence of AEs, by Action Taken With Regard to Study Medication
Description: Occurrence of AEs, by action taken with regard to study medication.
Time Frame: from day 1 and up to 4 weeks
Population: TS
Measure: Number; unit: percentage of participants
Groups:
- Treatment Naive (TN): Placebo: TN patient to receive Placebo +/- PegIFN/RBV for 28 days
- Treatment Experienced (TE) Non-cirrhotic: 48 mg QD: TE patient non-cirrhotic to receive 48mg QD solution BI201335 qd +/- PegIFN/RBV for 28 days
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants
  Action taken: decreasing dose | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.7 | 16.7 | 0.0
  Action taken: stop trial medication | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 28.6

17. Secondary Outcome: Occurrence of Discontinuations Due to AEs During BI201335 or BI201335+PegIFN/RBV Combination Treatment Period
Description: Occurrence of discontinuations due to AEs during BI201335 or BI201335+PegIFN/RBV combination treatment period.
Time Frame: from day 1 and up to 4 weeks
Population: TS
Measure: Number; unit: percentage of participants discontinued
Arm/Group | TN: Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
percentage of participants discontinued | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 28.6

18. Secondary Outcome: PK (Pharmacokinetic) Parameter After the First Dose: Cmax ( Maximum Measured Concentration of the Analyte in Plasma)
Description: PK (pharmacokinetic) parameter after the first dose: Cmax ( Maximum measured concentration of the analyte in plasma ).
  .
Time Frame: Times of -0:15, 0:30, 1:00, 2:00, 3:00, 4:00, 6:00. 8:00. 12:00, and 16:00 h relative to first administration of trial medication (on day 1)
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
ng/mL | 45.3 (53.9) | 170 (21.3) | 964 (66.1) | 2910 (51.6) | 164 (58.1) | 954 (30.5) | 2360 (48.3) | 7220 (48.8) | 7110 (86.8) | 5970 (162) | 7660 (68.1)

19. Secondary Outcome: PK Parameter After the First Dose: Tmax (Time From (Last) Dosing to the Maximum Measured Concentration of the Analyte in Plasma)
Description: PK parameter after the first dose: tmax (Time from (last) dosing to the maximum measured concentration of the analyte in plasma).
Time Frame: as for outcome 18
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
h | 7.07 (29.0) | 2.48 (149) | 2.12 (56.6) | 3.89 (44.1) | 3.89 (162) | 2.25 (59.1) | 3.23 (27.9) | 5.24 (49.2) | 5.30 (34.6) | 6.61 (14.9) | 5.63 (87.4)

20. Secondary Outcome: PK Parameter After the First Dose: AUCτ,1 (Area Under the Concentration-time Curve of the Analyte in Plasma Over a Uniform Dosing Interval τ on Day 1)
Description: PK parameter after the first dose: AUCτ,1 (Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ on day 1).
Time Frame: as for outcome 18
Population: TS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 7
ng*h/mL | 736 (57.0) | 2650 (16.5) | 11600 (52.9) | 35700 (48.2) | 2550 (48.3) | 12300 (47.5) | 27700 (59.9) | 108000 (55.5) | 52800 (82.6) | 78400 (157) | 56800 (55.7)

21. Secondary Outcome: PK Parameter at Steady State After the Last Dose: Cmax,ss (Maximum Measured Concentration of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: PK parameter at steady state after the last dose: Cmax,ss (Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ).
Time Frame: Times of -0:05, 0:30, 1:00, 2:00, 3:00, 4:00, 6:00. 8:00. 12:00, 16:00, 24:00 h relative to last administration of trial medication (on day 28)
Population: TS including patients with available Cmax,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
ng/mL | 150 (52.1) | 616 (62.4) | 4050 (43.3) | 15400 (40.4) | 478 (19.3) | 4170 (71.7) | 15400 (59.8) | 17700 (81.7) | 32200 (74.1) | 16400 (98.3) | 60400 (55.8)

22. Secondary Outcome: PK Parameter at Steady State After the Last Dose: Tmax,ss (Time From Last Dosing to the Maximum Measured Concentration of the Analyte in Plasma at Steady State )
Description: PK parameter at steady state after the last dose: tmax,ss (Time from last dosing to the maximum measured concentration of the analyte in plasma at steady state ).
Time Frame: as for outcome 21
Population: TS including patients with available tmax,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
h | 4.89 (52.0) | 3.38 (109) | 2.75 (27.6) | 3.36 (67.5) | 2.15 (45.5) | 1.94 (33.6) | 1.99 (46.7) | 3.23 (59.3) | 14.6 (14.1) | 4.12 (53.1) | 17.4 (18.2)

23. Secondary Outcome: PK Parameter at Steady State After the Last Dose: Cmin,ss (Minimum Measured Concentration of the Analyte in Plasma)
Description: PK parameter at steady state after the last dose: Cmin,ss (Minimum measured concentration of the analyte in plasma).
Time Frame: as for outcome 21
Population: TS including patients with available Cmin,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
ng/mL | 68.0 (52.4) | 199 (64.0) | 1120 (42.5) | 4040 (23.3) | 147 (43.6) | 863 (88.3) | 3640 (105) | 4970 (124) | 25500 (80.4) | 5870 (94.0) | 45400 (43.1)

24. Secondary Outcome: PK Parameter at Steady State After the Last Dose: AUCτ,ss (Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ)
Description: PK parameter at steady state after the last dose: AUCτ,ss ((Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ).
Time Frame: as for outcome 21
Population: TS including patients with available AUCτ,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 7 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
ng*h/mL | 2460 (53.9) | 8520 (55.6) | 49400 (42.8) | 185000 (21.1) | 6820 (22.1) | 43400 (75.9) | 164000 (83.8) | 221000 (82.2) | 350000 (75.6) | 243000 (75.8) | 642000 (46.1)

25. Secondary Outcome: PK Parameter at Steady State After the Last Dose: t1/2,ss (Terminal Half-life of the Analyte in Plasma at Steady State )
Description: PK parameter at steady state after the last dose: t1/2,ss (Terminal half-life of the analyte in plasma at steady state [h] )
Time Frame: as for outcome 21
Population: TS including patients with available t1/2,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
h | 30.5 (17.0) | 38.8 (41.2) | 25.5 (25.5) | 19.3 (12.4) | 33.2 (8.58) | 22.5 (17.4) | 22.1 (27.3) | 19.9 (25.0) | 27.3 (61.5) | 22.7 (33.0) | 41.5 (63.4)

26. Secondary Outcome: PK Parameter at Steady State After the Last Dose: MRTpo,ss (Mean Residence Time of the Analyte in the Body at Steady State After Oral Administration)
Description: PK parameter at steady state after the last dose: MRTpo,ss (Mean residence time of the analyte in the body at steady state after oral administration [h] )
Time Frame: as for outcome 21
Population: TS including patients with available MRTpo,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
h | 44.4 (17.0) | 60.2 (61.9) | 33.3 (23.5) | 26.7 (19.3) | 39.7 (14.0) | 26.6 (22.0) | 27.2 (37.4) | 30.7 (32.5) | 50.5 (59.9) | 34.2 (34.9) | 82.0 (71.6)

27. Secondary Outcome: PK Parameter at Steady State After the Last Dose: CL/F,ss (Apparent Clearance of the Analyte in Plasma at Steady State Following Multiple Oral Dose Administration )
Description: PK parameter at steady state after the last dose (if applicable): CL/F,ss (ss Apparent clearance of the analyte in plasma at steady state following multiple oral dose administration [mL/min] )
Time Frame: as for outcome 21
Population: TS including patients with available CL/F,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
mL/min | 136 (53.9) | 93.9 (55.6) | 40.4 (42.8) | 21.6 (21.1) | 117 (22.1) | 46.1 (75.9) | 24.4 (83.8) | 18.1 (82.2) | 11.4 (75.6) | 16.4 (75.8) | 6.23 (46.1)

28. Secondary Outcome: PK Parameter at Steady State After the Last Dose: Vz/F,ss (Apparent Volume of Distribution During the Terminal Phase z at Steady State Following an Oral Administration )
Description: PK parameter at steady state after the last dose: Vz/F,ss (Apparent volume of distribution during the terminal phase z at steady state following an oral administration [L] )
Time Frame: as for outcome 21
Population: TS including patients with available Vz/F,ss data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
L | 358 (46.7) | 315 (69.0) | 89.4 (34.1) | 36.1 (17.9) | 337 (26.7) | 89.9 (80.4) | 46.7 (65.3) | 31.0 (67.4) | 27.0 (54.4) | 32.3 (40.0) | 22.4 (27.1)

29. Secondary Outcome: PK Parameter for Drug-drug Interaction (naïve Patients With ≥1 Log Reduction on Day 10): AUCτ,ss (Area Under the Concentration-time Curve of the Analyte in Plasma at Steady State Over a Uniform Dosing Interval τ )
Description: PK parameter for drug-drug interaction (naïve patients with ≥1 log reduction on Day 10): AUCτ,ss ( Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ ).
Time Frame: Times of -0:05, 0:30, 1:00, 2:00, 3:00, 4:00, 6:00. 8:00. 12:00, 16:00, 24:00 h relative to administration of trial medication in the morning of Day 14 (on day 14)
Population: TS (for TN patients only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 6
ng*h/mL | 1970 (46.5) | 8740 (52.1) | 45800 (85.4) | 180000 (42.0)

30. Secondary Outcome: PK Parameter for Drug-drug Interaction (naïve Patients With ≥1 Log Reduction on Day 10): Cmax,ss
Description: PK parameter for drug-drug interaction (naïve patients with ≥1 log reduction on Day 10): Cmax,ss.
Time Frame: as for outcome 29
Population: TS (for TN patients only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 6
ng/mL | 106 (47.5) | 693 (61.1) | 3880 (82.8) | 13100 (38.2)

31. Secondary Outcome: PK Parameter for Drug-drug Interaction (naïve Patients With ≥1 Log Reduction on Day 10): Cmin, ss
Description: PK parameter for drug-drug interaction (naïve patients with ≥1 log reduction on Day 10): Cmin, ss.
Time Frame: as for outcome 29
Population: TS (for TN patients only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD
Number analyzed (Participants) | 6 | 7 | 6 | 6
ng/mL | 57.8 (46.2) | 185 (64.8) | 1010 (97.9) | 4320 (42.3)

32. Secondary Outcome: Accumulation Ratio of the Analyte in Plasma Following Multiple Doses Over a Uniform Dosing Interval: RAcmax
Description: For TN patients, comparing exposure on Day 14 to the first dose on Day 1; for TE patients, comparing exposure on Day 28 to the first dose on Day 1.
Time Frame: Day 1, Day 14, and Day 28
Population: TS including patients with available RAcmax data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
ratio | 2.34 (29.1) | 4.08 (66.6) | 3.74 (32.5) | 4.49 (36.2) | 2.91 (58.7) | 4.37 (50.6) | 6.53 (75.7) | 2.45 (89.4) | 4.53 (96.0) | 2.74 (90.5) | 6.81 (154)

33. Secondary Outcome: Accumulation Ratio of the Analyte in Plasma Following Multiple Doses Over a Uniform Dosing Interval: RAauc
Description: as for outcome 32
Time Frame: Day 1, Day 14, and Day 28
Population: TS including patients with available RAauc data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment Naive(TN): 20mg Per Day (QD) | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 7 | 6 | 15 | 15 | 6 | 5
ratio | 2.68 (19.6) | 3.30 (49.9) | 3.61 (42.0) | 5.03 (45.3) | 2.68 (36.2) | 3.52 (34.0) | 5.90 (56.6) | 2.05 (88.8) | 6.62 (88.8) | 3.11 (96.6) | 10.0 (111)

ADVERSE EVENTS:
Time Frame: day 1 and up to 4 weeks + washout
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive(TN): 20mg QD | TN: 48mg QD | TN: 120mg QD | TN: 240mg QD | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD | TE Non-cirrhotic: 120 mg QD | TE Non-cirrhotic: 240 mg QD | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) | TE Non-cirrhotic: 240 mg BID SGC | TE With Cirrhosis: 240 mg QD SGC | TE With Cirrhosis: 240 mg BID SGC
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/6 | 1/7 | 0/7 | 0/6 | 0/6 | 0/7 | 0/6 | 0/15 | 0/15 | 0/6 | 2/7
Other Adverse Events (participants affected / at risk) | 5/8 | 6/6 | 7/7 | 4/7 | 6/6 | 6/6 | 7/7 | 6/6 | 15/15 | 15/15 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (TN): Placebo (N=8) | Treatment Naive(TN): 20mg QD (N=6) | TN: 48mg QD (N=7) | TN: 120mg QD (N=7) | TN: 240mg QD (N=6) | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD (N=6) | TE Non-cirrhotic: 120 mg QD (N=7) | TE Non-cirrhotic: 240 mg QD (N=6) | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) (N=15) | TE Non-cirrhotic: 240 mg BID SGC (N=15) | TE With Cirrhosis: 240 mg QD SGC (N=6) | TE With Cirrhosis: 240 mg BID SGC (N=7)
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (TN): Placebo (N=8) | Treatment Naive(TN): 20mg QD (N=6) | TN: 48mg QD (N=7) | TN: 120mg QD (N=7) | TN: 240mg QD (N=6) | Treatment Experienced (TE) Non-cirrhotic: 48 mg QD (N=6) | TE Non-cirrhotic: 120 mg QD (N=7) | TE Non-cirrhotic: 240 mg QD (N=6) | TE Non-cirrhotic: 240 mg QD Soft Gel Capsule (SGC) (N=15) | TE Non-cirrhotic: 240 mg BID SGC (N=15) | TE With Cirrhosis: 240 mg QD SGC (N=6) | TE With Cirrhosis: 240 mg BID SGC (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 3 | 1 | 2 | 8 | 5 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 1 | 0 | 3 | 2 | 8 | 8 | 4 | 6
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 6 | 0 | 5
Asthenia (General disorders) | 2 | 3 | 3 | 0 | 4 | 1 | 2 | 1 | 3 | 5 | 2 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 4 | 2 | 4 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 3 | 11 | 3 | 3 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 3
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Mucosal ulceration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 2 | 4 | 2
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 6 | 2 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 3 | 0 | 3 | 2 | 2 | 3 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 2 | 1 | 2 | 2 | 3 | 3 | 9 | 10 | 4 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 5 | 2 | 3 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Larynx irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 3 | 0 | 3 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Photosensitivity allergic reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 2 | 4 | 1 | 3 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental implantation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.